CLINICAL TRIAL: NCT02621502
Title: Pilot Study to Evaluate the Glycemic Index, and the Satiating Effect Using Different Quinoa Varieties in a Group of Healthy Overweight Subjects
Brief Title: Quinoa Effects on Glycemic Index and Satiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Alicorp S.A.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: QUINOA
Record Dates: First submitted 2015-11-18; First posted 2015-12-03 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Overweight
Keywords: Quinoa; Satiety; Visual analogue scale; Cross-over studies
MeSH Terms: conditions — Overweight | interventions — Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Quinoa variety 1 (Experimental): 1 dose of Quinoa Variety 1 orally. The product is provided in a mix-pack together with water (100mL). This flexible container is capable of maintaining separate purified water (100 mL) and the experimental powder product in the same package. Both products can be easily mixed by breaking the inner seal. Volunteers had a maximum of 10 minutes to consume the product.
  Interventions: Dietary Supplement: Quinoa variety 1
- Quinoa variety 2 (Experimental): 1 dose of Quinoa Variety 2 orally. The product is provided in a mix-pack together with water (100mL). This flexible container is capable of maintaining separate purified water (100 mL) and the experimental powder product in the same package. Both products can be easily mixed by breaking the inner seal. Volunteers had a maximum of 10 minutes to consume the product.
  Interventions: Dietary Supplement: Quinoa variety 2
- Quinoa variety 3 (Experimental): 1 dose of Quinoa Variety 3 orally. The product is provided in a mix-pack together with water (100mL). This flexible container is capable of maintaining separate purified water (100 mL) and the experimental powder product in the same package. Both products can be easily mixed by breaking the inner seal. Volunteers had a maximum of 10 minutes to consume the product.
  Interventions: Dietary Supplement: Quinoa variety 3
- Quinoa variety 4 (Experimental): 1 dose of Quinoa Variety 4 orally. The product is provided in a mix-pack together with water (100mL). This flexible container is capable of maintaining separate purified water (100 mL) and the experimental powder product in the same package. Both products can be easily mixed by breaking the inner seal. Volunteers had a maximum of 10 minutes to consume the product.
  Interventions: Dietary Supplement: Quinoa variety 4
- Anhydrous Glucose (Active Comparator): 1 dose of Anhydrous Glucose orally. . The product is provided in a mix-pack together with water (100mL). This flexible container is capable of maintaining separate purified water (100 mL) and the control powder product in the same package. Both products can be easily mixed by breaking the inner seal. Volunteers had a maximum of 10 minutes to consume the product.
  Interventions: Dietary Supplement: Anhydrous Glucose

INTERVENTIONS:
Dietary Supplement: Quinoa variety 1 — On the intervention day, the volunteers will consume the Quinoa Variety 1.
  Then during minutes 0, 15, 30, 45, 60, 90, 120, 180, 240 and 260 two types of methodologies were conducted:
  * In minutes 0, 15, 30, 45, 60, 90 and 120, blood samples were collected.
  * In minutes 0, 15, 30, 60, 90, 120, 180, 240 and 260, volunteers completed the Visual analogue scale questionnaire.
  Arms: Quinoa variety 1
Dietary Supplement: Quinoa variety 2 — On the intervention day, the volunteers will consume the Quinoa Variety 2.
  Then during minutes 0, 15, 30, 45, 60, 90, 120, 180, 240 and 260 two types of methodologies were conducted:
  * In minutes 0, 15, 30, 45, 60, 90 and 120, blood samples were collected.
  * In minutes 0, 15, 30, 60, 90, 120, 180, 240 and 260, volunteers completed the Visual analogue scale questionnaire.
  Arms: Quinoa variety 2
Dietary Supplement: Quinoa variety 3 — On the intervention day, the volunteers will consume the Quinoa Variety 3.
  Then during minutes 0, 15, 30, 45, 60, 90, 120, 180, 240 and 260 two types of methodologies were conducted:
  * In minutes 0, 15, 30, 45, 60, 90 and 120, blood samples were collected.
  * In minutes 0, 15, 30, 60, 90, 120, 180, 240 and 260, volunteers completed the Visual analogue scale questionnaire.
  Arms: Quinoa variety 3
Dietary Supplement: Quinoa variety 4 — On the intervention day, the volunteers will consume the Quinoa Variety 4.
  Then during minutes 0, 15, 30, 45, 60, 90, 120, 180, 240 and 260 two types of methodologies were conducted:
  * In minutes 0, 15, 30, 45, 60, 90 and 120, blood samples were collected.
  * In minutes 0, 15, 30, 60, 90, 120, 180, 240 and 260, volunteers completed the Visual analogue scale questionnaire.
  Arms: Quinoa variety 4
Dietary Supplement: Anhydrous Glucose — On the intervention day, the volunteers will consume the control product.
  Then during minutes 0, 15, 30, 45, 60, 90, 120, 180, 240 and 260 two types of methodologies were conducted:
  * In minutes 0, 15, 30, 45, 60, 90 and 120, blood samples were collected.
  * In minutes 0, 15, 30, 60, 90, 120, 180, 240 and 260, volunteers completed the Visual analogue scale questionnaire.
  Arms: Anhydrous Glucose

SUMMARY:
The purpose of this study is to to assess the glycemic index and the satiating properties of different Quinoa varieties, using a Visual Analogue Scale in a sample of healthy overweight subjects.

DETAILED DESCRIPTION:
Pilot study to evaluate the glycemic index, and the satiating effect using different Quinoa varieties in a group of healthy overweight subjects.

ELIGIBILITY:
Inclusion Criteria:

* Men and women from 18 to 65 years old.
* Body mass index (BMI) ≥25 and <30 kg/m2.
* Adequate cultural level and understanding for the clinical trial.
* Signed informed consent

Exclusion Criteria:

* Individuals with BMI ≥30 or <25 kg/m2
* Vegetarians or individuals with a fiber intake ≥30 g/day
* Individuals diagnosed with Diabetes Mellitus
* Individuals with dyslipidemia on pharmacological treatment
* Individuals with hypertension on pharmacological treatment
* Smokers or heavy drinking individuals (>2-3 servings/day in men and > 1 serving/day in women (1 serving=1 glass of wine or 1 bottle of beer))
* Individuals with large weight fluctuations or who have undergone in recent months a weight loss diet
* Individuals with gastrointestinal diseases that affect the digestion or the absorption of nutrients
* Individuals receiving at least the preceding 2 months a pharmacological treatment that modifies the lipid profile (for example, statins, fibrates, diuretics, corticosteroids, oral antidiabetic medications)
* Pregnant or breastfeeding women
* Women with menstrual irregularities (absence of menstrual cycle at least 2 months prior)
* Individuals with intense physical activity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Glycemic index | 0, 15, 30, 45, 60, 90, 120 min
  The glycemic index is calculated with the incremental area under the curve of the glycemic response 7 time points ( 0 , 15 , 30, 45 , 60, 90 , 120 min) to 50 g intake carbohydrate food test food and reference

SECONDARY OUTCOMES:
Glucose metabolism related parameters | day 1, 8, 15, 22, 29
  glucose and insulin assessed in 7 point curves
satiety hunger assessment (visual analogue scale) | just before taking the product, just after taking the product, 30, 60 , 90, 120, 180, 240 min and 260 min after taking the product)
  visual analogue scale to assessment satiety and hunger will be picked up in 9 time points to calculate the area under the curve to get a score
Weight | day 1, 8, 15, 22, 29
  Weight
Adverse effects | day 1, 8, 15, 22, 29
  symptoms of gastrointestinal intolerance (nausea, diarrhea, bloating or other gastrointestinal disorder
Blood hormonal markers | just before taking the product, 15, 30, 45, 60, 90 and 120 min after consuming the product
  ghrelin, GLP-1 (glucagon-like peptide) and peptide YY
height | day 1, 8, 15, 22, 29
waist circumference | day 1, 8, 15, 22, 29
BMI | day 1, 8, 15, 22, 29
  body mass index

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Gómez Candela, MD, PhD, Principal Investigator — La Paz University Hospital
Locations (1):
- Hospital Universitairo La Paz, Madrid, Madrid, Spain

REFERENCES:
- See also: La Paz University Hospital Research Institute — http://www.idipaz.es/